CLINICAL TRIAL: NCT01114425
Title: Etude Observationnelle Multicentrique Relative à la tolérance de ISENTRESS® + TRUVADA® Prescrite en Prophylaxie Post-exposition de Personnes récemment Soumises au Risque de Transmission d'Une Infection Par le VIH
Brief Title: Safety Study of Isentress® + Truvada® in Post-exposure Treatment of HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Christian RABAUD, GERES
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 382426005_1
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
Keywords: tolerability of post exposure to HIV infection prophylaxis
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: raltegravir (Isentress) — raltegravir (Isentress) 400 mg bid
Drug: Truvada®

SUMMARY:
The objective are to assess the nature and incidence of drug intolerance observed with a new antiretroviral triple therapy, Truvada® [0-0-1] + Isentress® 400 mg tablets [1-0-1], prescribed in a setting of the treatment of individuals with recent exposure to a risk of transmission of HIV infection and to compare the results with those of previous studies conducted according to the same methodology, with other combinations of antiretrovirals.

ELIGIBILITY:
Inclusion criteria

* age 18 years or over
* consultation immediately following exposure to the risk of transmission of HIV infection (less than 48 hours, except in the case of rape when this period may be increased to a maximum of 120 hours)
* person capable of understanding the principle of the study and giving his/her informed consent

Exclusion criteria

* subjects recently exposed to a risk of transmission of HIV infection in which the source patient is known to be infected with HIV and treated, and whose therapeutic history justifies the introduction of PET other than that proposed in this study
* subjects with a contraindication to the prescription of Truvada® and/or Isentress® (renal impairment, allergy, etc.)
* subjects previously treated with phenytoin, phenobarbital and rifampicin, since combination with raltegravir is contraindicated subjects known to be infected with hepatitis B virus, whether or not treated with lamivudine
* subjects refusing to take part in the study
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
To assess the nature and incidence of drug intolerance and to compare the results with those of previous studies conducted according to the same methodology, with other combinations of antiretrovirals. | one year
  Proportion of patients who stop the post-exposure treatment before the planned 28 days, owing to adverse reaction(s).
  Proportion of patients reporting a post-exposure treatment-related side effect before the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian RABAUD, MD., PhD., Principal Investigator — Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux
Locations (1):
- GERES, Paris, France